CLINICAL TRIAL: NCT02634008
Title: An Open Label, Multicentre, International Pilot Study of Paritaprevir/Ritonavir, Ombitasvir, Dasabuvir With or Without Ribavirin or Glecaprevir/Pibrentasvir for People With Recently Acquired Hepatitis C Virus Infection With or Without HIV Co-infection.
Brief Title: Treatment of Recently Acquired Hepatitis C With the 3D Regimen or G/P
Acronym: TARGET3D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1502
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Hepatitis C, Acute
Keywords: Pangenotypic; Treatment
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; Viekira Pak; dasabuvir; Ribavirin; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Paritaprevir/ritonavir/ombitasvir (75mg/50mg/12.5mg) and dasabuvir (250mg) with or without ribavirin (1000-1200mg) daily taken orally for 8 weeks.
  Interventions: Drug: Paritaprevir/ritonavir/ombitasvir; Drug: Dasabuvir; Drug: Ribavirin
- Cohort 2 (Experimental): Three tablets of glecaprevir/pibrentasvir (100mg/40mg) daily taken orally for 6 weeks
  Interventions: Drug: Glecaprevir/pibrentasvir
- Cohort 3 (Experimental): Three tablets of glecaprevir/pibrentasvir (100mg/40mg) daily taken orally for 4 weeks
  Interventions: Drug: Glecaprevir/pibrentasvir

INTERVENTIONS:
Drug: Paritaprevir/ritonavir/ombitasvir
  Other Names: Viekira Pak
  Arms: Cohort 1
Drug: Dasabuvir
  Other Names: Viekira Pak
  Arms: Cohort 1
Drug: Ribavirin
  Arms: Cohort 1
Drug: Glecaprevir/pibrentasvir
  Arms: Cohort 2; Cohort 3

SUMMARY:
An open label, multicentre, international pilot study of paritaprevir/ritonavir, ombitasvir, dasabuvir with or without ribavirin or glecaprevir/pibrentasvir for people with recently acquired hepatitis C virus infection with or without HIV co-infection.

DETAILED DESCRIPTION:
The use of a highly potent IFN-sparing drug combination in the setting of recently acquired 1 HCV infection is hypothesised to result in the vast majority of patients achieving SVR. In this setting, it is anticipated that therapy can be shortened relative to that used in established chronic infection. A short course IFN-free strategy is likely to be highly attractive to both patients and clinicians and if proven may further encourage early HCV testing and diagnosis.

In this pilot study, the investigators plan to explore the safety, efficacy and feasibility of the IFN-sparing combination for treatment of recently acquired HCV infection.

Cohort One: paritaprevir/ritonavir/ombitasvir, dasabuvir with/without ribavirin (HCV genotype 1 only) Cohort Two (and Three): glecaprevir/pibrentasvir (HCV genotypes 1-6)

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent;
* Male and female patients aged 18 years and over;
* For Cohort One: willing to use two effective methods of contraception during the treatment period and 24 weeks post;
* For Cohort Two and Three: If female and of childbearing potential, willing to use at least one effective method of contraception during the treatment period and 4 weeks post; women not of childbearing potential include those who are postmenopausal or permanently surgically sterile (no contraception is required for male participants);
* For Cohort One, Two and Three: Females of child-bearing potential must have a negative pregnancy test at screening and immediately prior to first dose of study drugs;
* HCV genotype 1 infection at screening (Cohort 1 only);
* Detectable HCV RNA at screening (>10,000 IU/ml), and in the opinion of the investigator is unlikely to demonstrate spontaneous viral clearance;
* Absence of cirrhosis, as defined by one of the following:

  * Liver biopsy within 24 months prior to or during screening demonstrating absence of cirrhosis (eg, METAVIR fibrosis score ≤ 3, Ishak fibrosis score ≤ 4); or
  * FibroScan score < 12.5 kPa within ≤ 6 months of screening or during screening period; or
* Medically stable on the basis of physical examination, medical history and vital signs;
* Adequate English to provide reliable responses to the study questionnaires;
* Recently acquired HCV infection (estimated duration of infection ≤12 months) as defined by*:

  1. i) First anti-HCV Ab or HCV RNA positive within the previous 6 months and ii) Documented anti-HCV Ab negative within the 18 months prior to anti-HCV antibody positive result

     OR
  2. i) First anti-HCV Ab or HCV RNA positive within the previous 6 months and ii) Acute clinical hepatitis (jaundice or ALT> 10 X ULN) within the previous 12 months prior to first positive HCV antibody or HCV RNA, with no other cause of acute hepatitis identifiable

     OR
  3. i) First anti-HCV Ab or HCV RNA positive within the previous 6 months and ii) Acute asymptomatic hepatitis (acute rise in ALT> 5 X ULN) within the previous 12 months prior to first positive HCV antibody or HCV RNA and documented normal ALT within the previous 12 months with no othercause of acute hepatitis identifiable (In individuals with a previously high ALT, an acute rise to >3.5 x their previous peak ALT in last 12 months is acceptable)

     OR
  4. For cases of recent HCV reinfection the following criteria are required: Documented prior HCV antibody positive with HCV RNA negative on at least 2 occasions 6 months apart AND new HCV RNA positive within the previous 6 months.

     * Estimated duration of infection based on midpoint between last antibody or RNA negative and first antibody or HCV RNA positive in the case of seroconversion and 6 weeks prior to date of maximum ALT in the case of acute hepatitis.

     If co-infection with HIV is documented, the subject must meet the following criteria:

     Cohort One:
* On a stable qualifying ARV regimen for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and a plasma HIV RNA below the limit of detection.

Cohort Two:

• On a stable qualifying ARV regimen for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and a plasma HIV RNA below the limit of detection.

OR

• ARV naïve with CD4 T cell count >500 cells/mm3

Exclusion Criteria:

* Pregnancy/lactation
* Infection or co-infection with an HCV genotype other than 1 (Cohort 1 only)
* Subject has current or past clinical evidence of decompensated liver disease, such as ascites, hepatic encephalopathy, oesophageal varices, and/or any of the following screening laboratory results;

  * International Normalized Ration (INR) > 1.5;
  * Patients with a known inherited blood disorder and INR > 1.5 may be enrolled after discussion with the Principal Investigator
  * Serum albumin <3.3 g/dL;
  * Serum total bilirubin >1.8 x upper limit of normal (ULN), unless isolated in subjects with Gilbert's syndrome;
* Subject shows evidence of significant liver disease in addition to hepatitis C, which may include but is not limited to drug- or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, non-alcoholic steatohepatitis (NASH), or primary biliary cirrhosis;
* Subject has active malignant disease or history of malignant disease within the past 5 years (with the exception of treated basal cell carcinoma);
* History of chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study;
* Poorly controlled diabetes mellitus as evidenced by haemoglobin A1c (HbA1c) ≥8.5%;
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤6 months prior to the first dose of study drug
* Prior treatment failure with an HCV protease inhibitor;
* Any investigational drug ≤6 weeks prior to the first dose of study drug;
* Positive test at screening for anti-HAV IgM Ab, anti-HBc IgM Ab or HBsAg;
* Confirmed presence of hepatocellular carcinoma indicated on imaging techniques such as computed tomography (CT) scan or magnetic resonance imaging (MRI) within 3 months prior to screening or on an ultrasound performed at screening (a positive ultrasound result will be confirmed with CT scan or MRI);
* Subject has history of organ transplant that requires chronic immunosuppression

  * Corneal, skin, and hair grafts are allowed;
* History of severe psychiatric disease that in the opinion of the investigator is unstable enough to compromise treatment adherence;
* Subject has evidence of serious or severe bacterial or fungal infection(s), including active tuberculosis;
* Prohibited medications and herbal remedies as detailed in section 5.5;
* Screening laboratory tests showing any of the following abnormal results:

  * Haemoglobin <100 g/L
  * Calculated creatinine clearance <50mL/min
  * Platelets <100,000 cells/mm3
  * Absolute neutrophil count (ANC) <1,500 cells/µL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of treated subjects (intention-to-treat (ITT) population) demonstrating undetectable hepatitis C virus (HCV) RNA at 12 weeks following treatment (SVR 12). | 12 weeks post treatment

SECONDARY OUTCOMES:
The proportion of treated subjects overall with ETR, SVR4 and SVR24 defined as undetectable HCV RNA at end of therapy, 4 weeks and 24 weeks post therapy, respectively. | End of treatment- week 6 or week 8 depending on the study arm; 4 weeks post treatment; 24 weeks post treatment
Comparison of ETR, SVR4, SVR12 and SVR24 between those receiving 8 weeks treatment and those receiving 6 weeks treatment. | End of treatment- week 6 or week 8 depending on the study arm; 4 weeks post treatment; 12 weeks post treatment; 24 weeks post treatment
Comparison of adherence between those receiving 8 weeks treatment and those receiving 6 weeks treatment | Baseline to week 6 or week 8 treatment duration
Proportion with early treatment discontinuation | Baseline through to 6 or 8 weeks depending on the study arm
Proportion with adverse events (including serious adverse events) | Baseline to week 6 or week 8 treatment duration
Changes in laboratory parameters, including liver function tests (ALT, AST) and haematological indices (haemoglobin, neutrophil count, platelet count) | Baseline to week 6 or week 8 treatment duration
Emergence of resistance associated variants (RAVs) | Baseline through to 6 or 8 weeks depending on the study arm
HCV reinfection rate | Week 208
Changes in sexual and injecting drug use behaviour at SVR 12 and end of follow up | 12 weeks post treatment; week 208
Serum cytokine and ISG expression at baseline and week 4 | Baseline; week 4 on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MBBS PhD, Principal Investigator — Kirby Institute
Locations (11):
- Australia (3):
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
- New Zealand (2):
  - Auckland City Hospital, Auckland, Grafton
  - Christchurch Hospital, Christchurch
- United Kingdom (6):
  - Barts and London, London
  - Royal Free Hospital, London
  - Guy's and St Thomas' Hospital, London
  - Chelsea and Westminster Hospital, London
  - St Mary's Hospital, London
  - Pennine Acute Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinello M, Bhagani S, Shaw D, Orkin C, Cooke G, Gane E, Iser D, Ustianowski A, Kulasegaram R, Stedman C, Tu E, Grebely J, Dore GJ, Nelson M, Matthews GV. Glecaprevir-pibrentasvir for 4 weeks among people with recent HCV infection: The TARGET3D study. JHEP Rep. 2023 Jul 27;5(10):100867. doi: 10.1016/j.jhepr.2023.100867. eCollection 2023 Oct. PMID 37771545